CLINICAL TRIAL: NCT03848234
Title: A Randomized Trial Administering Estradiol Patch vs. Placebo Patch as add-on to Antipsychotics in Patients With Schizophrenia, Schizoaffective or Schizophreniform Disorder
Brief Title: Estradiol Patch as add-on to Antipsychotics in Patients With Schizophrenia, Schizoaffective or Schizophreniform Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tangent Data (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EST-S-01
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Randomized, add-on to anti-psychotics, double blind, placebo-controlled, parallel group clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Estradiol (Experimental): 2 trans dermal patches to be changed twice a week for the duration of 8 weeks
  Interventions: Drug: Estradiol; Device: Placebo
- B Placebo (Placebo Comparator): 2 trans dermal patches to be changed twice a week for the duration of 8 weeks
  Interventions: Drug: Estradiol; Device: Placebo

INTERVENTIONS:
Drug: Estradiol — 2 trans dermal patches to be changed twice a week for the duration of 8 weeks.
  Other Names: trans dermal patches
Device: Placebo — 2 trans dermal patches to be changed twice a week for the duration of 8 weeks.
  Other Names: trans dermal patches

SUMMARY:
To evaluate the effects of Estradiol patches vs placebo patches as add-on to antipsychotics on psychometric performance in patients with schizophrenia, schizoaffective or schizophreniform disorder

DETAILED DESCRIPTION:
Estradiol has been shown to be an effective adjunctive treatment for schizophrenia. The estradiol hypothesis was tested in a randomized-controlled trial in which estradiol was given to women with schizophrenia, schizoaffective or schizophreniform disorder aged 18 to 45 - Kulkarni 2014. In that 3 arms trial, Kulkarni administered transdermal 100 µg estradiol/200 µg estradiol/ placebo to patients receiving anti-psychotics and reported reductions in PANSS positive, general and total symptoms in both estradiol patients' groups compared with the placebo group. Patients receiving 200 µg experienced greater improvement, specifically in the PANSS positive subscale, the effect size was 0.44.

The objective of this study is to attempt to confirm Kulkarni's trial in a large-scale trial. This proposed study is a 2-arm study, in which patients will be randomized to either 200 µg estradiol or placebo in order to test the effectiveness of estradiol on women of childbearing age with schizophrenia, schizoaffective or schizophreniform disorder for a limited period of 56 days.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18-45 years of age, inclusive
2. Willing and able to provide informed consent, after the nature of the study has been fully explained
3. Current DSM-IV-TR diagnosis of schizophrenia, schizoaffective or schizophreniform disorder as confirmed by modified SCID.
4. Total PANSS score > 60 and (PANSS positive subscale >15 and/or PANSS negative subscale >15)
5. Must be on a stable dose of any antipsychotic drug, for at least 2 weeks prior to the baseline visit, at doses within the PORT criteria, whenever possible. Patients receiving higher doses will have their records reviewed to insure that their dose is required and, if possible, will be stabilized on a lower dose prior to study entry.
6. Patients who are physically and endocrinologically healthy,
7. Inpatients or outpatients. Inpatients will be randomized 3 days or more after admission

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Pregnant or breast-feeding
3. Women who are menopausal.
4. Patients treated with oral estrogen preparations containing estradiol greater than 30 mcg.
5. Women who have known severe abnormalities in the hypothalamo-pituitary gonadal axis, thyroid disorders, severe medical conditions and disorders that would contraindicate estrogen use (breast cancer, migraine with aura or stroke)
6. History of endometrial cancer or breast cancer, vaginal bleeding between periods, untreated endometrial hyperplasia, previous or present thrombembolism, known thrombophilic disorders, abnormal liver function tests, porphyria.
7. History of 1st and 2nd grade family with breast or uterine cancer,
8. Likely allergy or sensitivity to estradiol.
9. Schizoaffective disorder in the manic phase.
10. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
11. Patients with a current DSM-IV substance or alcohol abuse. Patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
12. Concurrent delirium, mental retardation, drug-induced psychosis, or history of clinically significant brain trauma documented by CT or MRI.
13. Patients receiving phenobarbital, phenytoin, carbamazepine, rifampicin, rifabutin, nevirapine, efavirenz, ritonavir and nelfinavir,or Hypericum perforatum

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 209 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
PANSS positive subscale at the end of the trial | 8 weeks
  To evaluate the effects of Estradiol on Positive and Negative Syndrome Scale for Schizophrenia (PANSS)

SECONDARY OUTCOMES:
PANSS total, negative and general psychopathology scales | 8 weeks
  To evaluate the effects of Estradiol on Positive and Negative Syndrome Scale for Schizophrenia (PANSS)
Clinical Global Impression Scale-Severity (CGI-S) and Global Impression Scale-Improvement (CGI-I) | 8 weeks
  To evaluate the effects of Estradiol on Clinical Global Impression
Brief Assessment of Cognition in Schizophrenia (BACS), | 8 weeks
  To evaluate the effects of Estradiol on cognition
Montgomery-Asberg Depression Rating Scale | 8 weeks
  To evaluate the effects of Estradiol on depressive symptoms
Rates of drop outs before the end of the trial | through study completion, an average of 1 year
  To evaluate the rate of drop outs

CONTACTS AND LOCATIONS:
Overall Officials: Paull G Radu, M.D., Study Director — Tangent Data
Locations (1):
- Clinical Psychiatric Hospital, Codru, Chișinău Municipality, Moldova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weiser M, Levi L, Zamora D, Biegon A, SanGiovanni JP, Davidson M, Burshtein S, Gonen I, Radu P, Slobozean Pavalache K, Nastas I, Hemi R, Ryan T, Davis JM. Effect of Adjunctive Estradiol on Schizophrenia Among Women of Childbearing Age: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Oct 1;76(10):1009-1017. doi: 10.1001/jamapsychiatry.2019.1842. PMID 31365044